CLINICAL TRIAL: NCT00882102
Title: Phase II Study of Decitabine and Gemtuzumab Ozogamicin in Acute Myelogenous Leukemia and High-Risk Myelodysplastic Syndrome
Brief Title: Decitabine and Gemtuzumab Ozogamicin in Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (H-R MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0288
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myelogenous Leukemia; High-Risk Myelodysplastic Syndrome; AML; MDS; Leukemia; Decitabine; Gemtuzumab Ozogamicin; Dacogen; Mylotarg
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Decitabine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine + Gemtuzumab Ozogamicin (Experimental): Decitabine 20 mg/m^2 by vein (IV) over 1-1/2 hours daily for 5 days. Gemtuzumab ozogamicin 3 mg/m^2 by vein on day 5.
  Interventions: Drug: Decitabine; Drug: Gemtuzumab ozogamicin

INTERVENTIONS:
Drug: Decitabine — Decitabine 20 mg/m^2 IV over 1-1/2 hours daily for 5 days.
  Other Names: Dacogen®
Drug: Gemtuzumab ozogamicin — Gemtuzumab ozogamicin 3 mg/m^2 IV on day 5.
  Other Names: Mylotarg®

SUMMARY:
The goal of this clinical research study is to learn if 5-aza-2 deoxycytidine (decitabine) given in combination with Mylotarg (gemtuzumab ozogamicin) can help to control Acute myeloid leukemia (AML), high-risk myelodysplastic syndromes (MDS) or Myelofibrosis (MF). The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Gemtuzumab ozogamicin is designed to attach to Sialic acid-binding Ig-like lectin 3 (CD33), a certain protein that is often found in leukemia cells, causing them to die.

Decitabine is designed to damage the Deoxyribonucleic acid (DNA) (the genetic material) of cells, which may cause cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive decitabine through a needle in your vein over 1 and 1/2 hours on Days 1-5 of each cycle. You will also receive gemtuzumab ozogamicin by vein over about 1 hour after you receive decitabine on Day 5 of each 4-8 week cycle.

During Cycle 1 only, if a bone marrow test done 2 weeks after you receive your first study drug treatment shows abnormal leukemia cells, you will receive another treatment with decitabine by vein over 1 and 1/2 hours for 5 days.

Gemtuzumab may cause allergic reactions, nausea, and vomiting. To help decrease the risk of such side effects, you will receive Benadryl (diphenhydramine), acetaminophen, meperidine, and hydrocortisone. You may receive these drugs by vein, or by mouth on each of the days you get gemtuzumab ozogamicin.

Study Visits:

At every study visit, you will be asked if you have experienced side effects and to list any drugs you may be taking.

During Cycle 1, blood (about 2 teaspoons) will be drawn at least 1 time each week for routine tests. If the doctor thinks it is necessary, you may be asked to have additional blood drawn.

On Day 1 of every cycle, your performance status will be recorded and your vital signs will be measured.

On Days 1-5 of Cycle 1, your vital signs will be measured.

Between Days 12 and 16 of Cycle 1, you will have a bone marrow aspirate if you have a diagnosis of AML or high-risk MDS to check the status of the disease. This test may be delayed if your doctor does not think you are in remission.

During Cycles 2-3, blood (about 2 teaspoons) will be drawn for routine tests at least 2 times each month.

On Day 1 of Cycles 2 and beyond, you will have a physical exam, including measurement of your vital signs.

During Cycles 4 and beyond, blood (about 2 teaspoons) will be drawn for routine tests at least 1 time each month.

If the doctor thinks it is necessary, you will have a bone marrow aspirate every 1-3 months to check the status of the disease.

You should tell the study doctor about all drugs and supplements you are taking while you are on this study.

Length of Study:

You may receive the combination of decitabine and gemtuzumab ozogamicin for up to 6 cycles. After this, if your doctor thinks it is in your best interest, you may continue to receive decitabine alone for up to 24 cycles. During this part of study, your performance status will be recorded, you will have a physical exam, and your vital signs will be measured on Day 1 of each cycle. Blood (about 2 teaspoons) will be drawn for tests once a month. You will be taken off study early if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to receive the study drug(s).

Long-Term Follow-up:

Once you are off study, you will have follow-up visits every month for up to 2 years. At these visits, blood (about 2 teaspoons) will be drawn for routine tests.

This is an investigational study. Gemtuzumab ozogamicin is FDA approved and commercially available for the treatment of AML that has come back after treatment in patients over the age of 65 years. Decitabine is FDA approved and commercially available for the treatment of MDS. The use of gemtuzumab ozogamicin and decitabine in combination is investigational.

Up to 100 participants will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >/= to 16 years at the time of signing the informed consent form.
3. Diagnosis of AML [other than acute promyelocytic leukemia (APL)] with refractory/relapsed disease. Patients with newly diagnosed AML will be eligible if not a candidate for intensive chemotherapy. Patients with high-risk (intermediate-2 or high by International Prognostic Scoring System (IPSS) or >/= 10% blasts) MDS will also be eligible. All non-hematological toxicity of previous cancer therapy should have resolved to </= grade 1 (except alopecia or other toxicities not involving major organs).
4. Eastern Cooperative Oncology Group (ECOG) performance status of </=3 at study entry.
5. Laboratory test results within these ranges (unless due to leukemia): Serum creatinine </= 2 mg/dL Total bilirubin </= 2 mg/dL aspartate aminotransferase (AST) (SGOT) and/or alanine aminotransferase (ALT) (SGPT) </= 2.5 * upper limit of normal (ULN) or </= 5 * ULN if related to disease
6. Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 days and must either commit to continued abstinence from heterosexual intercourse or adopting at least one highly effective method of contraception. These methods include intra-uterine device, tubal ligation, partner's vasectomy, hormonal birth control pills. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.
7. Active participants of the similar Protocol 2007-0882 (preceding study of decitabine and Mylotarg) are eligible to roll-over to this protocol without meeting the inclusion or exclusion criteria for this study.
8. For patients with MF only: Diagnosis of MF requiring therapy, including those previously treated by MF-directed therapy and relapsed or refractory; or if newly diagnosed then with intermediate or high risk according to Lille scoring system (adverse prognostic factors are: hemoglobin (Hb) < 10 g/dl, White blood cells (WBC) < 4 or > 30 * 10^9/L; risk group: 0 = low, 1 = intermediate, 2 = high), or with symptomatic splenomegaly (>/=10cm below left mid-costal margin).
9. For patients with MF only: Performance status 0-2 (Zubrod).
10. For patients with MF only: Signed informed consent.
11. For patients with MF only: Patients must have been off MF-directed therapy for 2 weeks prior to entering this study and have recovered from the toxic effects (grade 0-1) of that therapy. Patients are allowed to enter the study if on stable dose, for at least 1 months, of anagrelide (to control high platelets) or hydroxyurea (to control high WBC or enlarging spleen), or on stable dose, for at least 2 months, of erythropoietin (for significant anemia).
12. For patients with MF only: Serum bilirubin levels </= 2 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis, as judged by treating physician.
13. For patients with MF only: Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels </= 2* ULN, unless related to the MF, as judged by treating physician.
14. For patients with MF only: Serum creatinine levels </= 2* ULN.
15. For patients with MF only: Women of childbearing potential must have a negative serum pregnancy test prior to treatment and should be advised to avoid becoming pregnant. Men must be advised to not father a child while receiving treatment. Both women of childbearing potential and men must practice effective methods of contraception (those generally accepted as standard of care measures).
16. For patients with MF only: Age > 18 years.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk.
3. Use of any other experimental drug or therapy for leukemia within 14 days unless there is clear evidence of rapid disease progression. Use of hydrea to control proliferative disease will be allowed prior to starting therapy on study and for up to 7 days each during cycle 1-3 (Maximum daily dose of 7 gm).
4. For patients with MF only: Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
5. For patients with MF only: Uncontrolled intercurrent illness including, but not limited to, uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center's official website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 04/02/09 through 6/23/2010. All participants recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the forty-three participants registered only forty participants received treatment and were evaluable for toxicity and response.
Groups:
- Decitabine + Gemtuzumab Ozogamicin: Decitabine 20 mg/m2 by vein over 1-1/2 hours daily x 5. Gemtuzumab ozogamicin 3 mg/m2 by vein on day 5.
Period: Overall Study
Arm/Group | Decitabine + Gemtuzumab Ozogamicin
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 40
Age Continuous [Median (Full Range); unit: years] | 74 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response
Description: Complete Response (CR) was defined as normalization of peripheral blood and bone marrow with </= 5% blasts, a peripheral absolute neutrophil count (ANC) >/= 1 * 10^9 /l, and a platelet count of >/= 100 & 10^9 /l. Approximately Day 14 of the first cycle of 4 - 8 week cycle, a bone marrow aspirate was performed to check the status of the disease using International Working Group (IWG) criteria for acute myelogenous leukemia (AML) and myelofibrosis (MF).
Time Frame: Day 14 of first cycle
Measure: Number; unit: Participants
Groups:
- Decitabine + Gemtuzumab Ozogamicin: Decitabine 20 mg/m^2 by vein over 1-1/2 hours daily for 5 days. Gemtuzumab ozogamicin 3 mg/m^2 by vein on day 5.
Arm/Group | Decitabine + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 40
Participants | 10

ADVERSE EVENTS:
Time Frame: Three years, four months.
Arm/Group | Decitabine + Gemtuzumab Ozogamicin
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Gemtuzumab Ozogamicin (N=40)
Elevated Amylase/Lipase (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Gemtuzumab Ozogamicin (N=40)
Hemorhage (Gastrointestinal disorders) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 20 (20)
Infection (Infections and infestations) | 4 (4)
Mucositis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes